CLINICAL TRIAL: NCT04425525
Title: Adaptation of The Functional Difficulties Questionnaire-shortened Version Survey to Turkish and Determination of Psychometric Properties: Validity and Reliability Study.
Brief Title: The Functional Difficulties Questionnaire-shortened Version: Turkish Translation, Validity and Reliability Study.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Muğla Sıtkı Koçman University (Other)
Collaborators: Aydın Private Medinova Hospital (Unknown)
Responsible Party: Principal Investigator, Ayşe Adıgüzel Bayar, Physiotherapist, Muğla Sıtkı Koçman University
Other Study IDs: MSc Thesis
Record Dates: First submitted 2020-06-04; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Functional Status After CABG Surgery; Outcome Measure
Keywords: heart surgery, function, measure, validity, reliability.

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 15 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Functional Difficulties Questionnaire-shortened version "(FDQ-s) is a unique questionnaire that aimed at evaluating the functional performance of the upper extremities and trunk following cardiothoracic surgery.

Aim of this study is adaptation of the FDQ-s questionnaire to Turkish culture and study its psychometric properties, validity and reliability.

DETAILED DESCRIPTION:
Cardiac surgeries performed by sternotomy method are the most common surgical treatment method in coronary artery disease. Although the median sternotomy has advantages in terms of ease of application, cost and long-term survival, muskuloskeletal complications can be encountered in the postoperative period.

In the studies conducted, it was found that patients had difficulties in functional activities including mobilization and daily life activities after median sternotomy. Also restrictions or loss of motion can be observed in the joint range of motion of the shoulder joint and thoracic region.

The FDQ-s scale consists of 10 functional tasks developed by Sturgess et al. These tasks are activities such as coughing, sneezing, deep breathing, movements involving the upper extremity, turning in bed, sitting upright in the chair, and ambulation. When applying FDQ-s, patients will mark how hard they are in each task on the 100 mm straight line. The first point on the left means "no difficulty" and the last point on the right means "maximum difficulty". The score will be determined by measuring from the starting point to the place marked by the patient. The total score is at most 100 points and at least 0 points. The high score indicates that the patient's difficulty level is high.

Although there are many functional difficulties faced by patients in the postoperative period, there is no outcome measurement in our language that evaluates the level of these difficulties globally and objectively.

Our research will be done due to the elimination of this deficiency in the literature.

ELIGIBILITY:
Inclusion Criteria:

* Being over the age of 18
* Having undergone coronary artery bypass surgery (via median sternotomi)

Exclusion Criteria:

* Not having ability to read and write in Turkish
* Having cognitive impairment
* Being in the intensive care unit for more than five days due to medical reasons.
* Having undergone surgery involving thorax or upper extremity in the last 6 months.
* Having neurologic or musculoskeletal problems to prevent evaluation, ambulation and exercise.
* Patients who have an infection or unhealed scar after surgery even if their first measurements are made

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Having undergone coronary artery bypass surgery with median sternotomi
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-06-18 (Estimated)

PRIMARY OUTCOMES:
Change of the Functional Status (with FDQ-s: Turkish version questionnaire) | First day at the hospital (pre-op), day of discharge (post-op), 15th day after surgery (control).
  FDQ-S is a questionnaire created to evaluate the difficulties faced by patients undergoing cardiac surgery, especially when performing functional tasks of the thoracic region and upper extremity. The questionnaire consisting of 10 questions in total, the patients marked how much difficulty they had in each task, on a 100 mm straight line.The first point on the left means "no difficulty" and the last point on the right means "maximum difficulty". The score was determined by measuring from the starting point to the place marked by the patient. The total score is at most 100 points and at least 0 points. The high score indicates that the patient's strain level is high. With time frames we aimed to evaluate the change of the difficulty of patients function.

SECONDARY OUTCOMES:
Change of the Mobility Status : (Barthel İndex of Activities of Daily Living) | Day of discharge (post-op), 15th day after surgery (control day).
  Barthel Index determines the level of addiction of the patient in 10 sections: nutrition, washing, self-care, dressing and bowel care, bladder care, toilet care, wheelchair to bed and vice versa, mobility (walking on a smooth surface, using the wheelchair: if appropriate), going up and down stairs.The total score is in the range of 0-100, which means 0-20 points: fully dependent, 21-61: highly dependent, 62-90: moderately dependent, 91-99: slightly dependent, 100 points: fully independent.With time frames we aimed to evaluate the change of the mobility scores.
Change of the Quality of Life Status: (SF-36 Quality of Life Questionnaire) | Day of discharge (post-op), 15th day after surgery (control day).
  SF-36 is the most common scale used to measure individuals' quality of life. This scale examines 8 dimensions of health with 36 items such as physical function, role restrictions (due to physical and emotional problems), social function, mental health, vitality (energy), pain and general perception of health.Instead of giving only one total score, the scale gives total score separately for each subscale.100 points indicate good health, 0 points indicate bad health. With time frame we aimed to evaluate the cange of the life quality score of patients.
Change of the Pain Status: (Visual Analogue Scale) | First day at the hospital (pre-op), day of discharge (post-op), 15th day after surgery (control day).
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain." The distance from the 0 point to the place marked by the patient indicates the pain of the patient. With time frame we aimed to evaluate the change of the life quality score of patients.
Change of the Mobility Status: (Perme Intensive Care Mobility Score) | Day of discharge (post-op), 15th day after surgery (control day).
  The Perme ICU Mobility Score is a tool developed to measure the patient's mobility status starting with the ability to follow commands and culminating in the distance walked in two minutes. A total score of 3 or 4 is given for each item, reflecting the patient's mobility. A high score indicates a small amount of mobility barrier and low help, while a low score indicates more mobility and more help needed for mobility. With time frame we aimed to evaluate the change of the mobility score.

OTHER OUTCOMES:
Age | First day at the hospital (pre-op)
  Age (Year)
Height | First day at the hospital (pre-op)
  Height in meters
BMI | First day at the hospital
  BMI (weight and height combined to report BMI in kg/m²)

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Adıgüzel Bayar, MSc Student, Principal Investigator — Muğla Sıtkı Koçman University/ Private Medinova Hospital; Baki Umut Tuğay, Prof. Dr., Study Director — Muğla Sıtkı Koçman University
Locations (1):
- Private Medinova Hospital, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided